CLINICAL TRIAL: NCT06551701
Title: A Cluster-randomized Trial to Improve Use of High IntEnsity Statins for Vascular Protection
Brief Title: ACHIEVE Pilot Statins for Vascular Protection
Acronym: ACHIEVE
Status: Active, not recruiting | Type: Observational
Sponsor: Duke University (Other)
Collaborators: Carelon Research (Other); Harvard Pilgrim Health Care (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: Pro00114111; 1R34HL166680-01A1 (NIH)
Record Dates: First submitted 2024-08-05; First posted 2024-08-13 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: ASCVD
Keywords: Statin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- No statin: Patients who are identified with ASCVD who do not take a statin or do not take the recommended dose.
  Interventions: Other: Pharmacist call

INTERVENTIONS:
Other: Pharmacist call — Pharmacists will call patients and their providers to discuss benefits of statin use

SUMMARY:
ACHIEVE aims to increase statin usage among patients with ASCVD by having a pharmacist talk to patients and providers.

DETAILED DESCRIPTION:
Atherosclerotic cardiovascular disease (ASCVD) is the leading cause of death in the United States (U.S.) Statins reduce the risk of cardiovascular events by 30% in those with prior history of ASCVD. Despite being inexpensive and well-tolerated, however, statins are underused in clinical practice, particularly in patients who identify as Black. A large-scale intervention to improve evidence-based statin initiation among individuals with ASCVD is needed, particularly for the Black population. To meet this need, we aim to conduct a multi-center, pragmatic, cluster randomized, controlled trial to assess the impact of a provider- and patient-directed intervention to increase the prescription of, and adherence to, appropriate statin therapy among those with ASCVD (ACHIEVE: A Controlled trial to improve use of High IntEnsity statins for Vascular protEction). The intervention will be pharmacist-led, embedded in commercial payer systems, partnering with the National Committee for Quality Assurance (NCQA), and with a particular emphasis on improving statin use in the Black population.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of atherosclerotic cardiovascular disease currently not treated with a moderate- high intensity statin and the providers that care for them.
* Patient age 18-75

Exclusion Criteria:

* Hemodialysis
* History of rhabdomyolysis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes patients who have an ASCVD diagnosis but are currently not treated with a moderate-high intensity statin.
Sampling Method: Non-Probability Sample
Enrollment: 225 (Actual)
Dates: Start 2025-05-19 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Provider engagement as measured by recruitment | 2 years
  The goal is recruiting at least 25% of identified providers.
Patient engagement as measured by recruitment | 2 years
  The goal is to recruit at least 30% of identified patients overall and within the black population

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Granger, MD, Principal Investigator — Duke University
Locations (2):
- United States (2):
  - Carelon Research, Wilmington, Delaware
  - Duke Clinical Research Institute, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
We will provide requested unrestricted data to parties who sign a data sharing agreement which stipulates that data must be: 1) used solely for research purposes, 2) properly acknowledged in resulting publications, 3) kept confidential and inaccessible to third parties, and 4) destroyed or returned after analyses are completed. Additionally, users must agree not to use data to identify individual participants. Letters of agreement will be executed so that research materials can be provided to not-for-profit institutions. The study team further agrees that all resource sharing agreements comply with the Bayh-Dole Act of 1980 and the Technology Transfer Commercialization Act of 2000. We will not be using model organisms.
Supporting Information: Study Protocol
Time Frame: Data will be shared after publication of the final manuscript and will continue until the data from the main study is available for sharing.
Access Criteria: Unrestricted access will be provided to parties who sign a standard data sharing agreement.